CLINICAL TRIAL: NCT04992845
Title: Fusionless Treatment of Idiopathic Scoliosis With the SCOLI-TETHER System During The Growth Period
Acronym: FUTURE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Sponsor decided to focus their resources on the clinical data collection for the second generation of the investigational device.
Sponsor: Spino Modulation Inc. (Industry)
Responsible Party: Sponsor
Organization: Spinologics Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD-0001-PRO
Record Dates: First submitted 2021-07-23; First posted 2021-08-05 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-04

CONDITIONS: Adolescent Idiopathic Scoliosis; Juvenile Idiopathic Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Vertebral Body Tethering surgery
  Interventions: Device: Anterior Vertebral Body Tethering

INTERVENTIONS:
Device: Anterior Vertebral Body Tethering — The SCOLI-TETHER (MIScoli) System is intended for anterolateral vertebral body fixation and internal fastening of the convex side of the thoracic curvatures thereby reducing the deformity and preventing the progression of idiopathic scoliosis in growing children/adolescents at high risk for curve progression while preserving motion.

SUMMARY:
The goal of the study is to establish the safety and benefit of treatment of juvenile and adolescent idiopathic scoliosis (AIS) with the SCOLI-TETHER (MIScoli) System.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of juvenile or adolescent idiopathic scoliosis
2. Male and female subjects greater than 8 years of age with significant growth remaining
3. Risser Stage 0 or 1
4. Subjects should have at least three years of estimated growth remaining based on Risser staging
5. Major thoracic scoliosis with Cobb Angle > 40° and < 70° and Lenke I, II or V curve pattern. Cobb measurements refer to measures taken without a brace. Patients with curves greater than 30 degrees with attempted but failed brace treatment are also potential candidates for the procedure
6. Thoracic kyphosis (T5-T12) < 50°
7. Instrumentation to be applied no more cephalad than T4 and no more caudal than L2 (inclusive)
8. Menses < 4 months
9. Subject must be physically and mentally willing and able to comply with postoperative and routinely scheduled clinical and radiographic evaluations
10. Subject assent and parent/legal guardian consent obtained and documented.

Exclusion Criteria:

1. Scoliosis curve is less than 30° or more than 70°
2. Thoracic kyphosis is greater than or equal to 50° (T5-T12)
3. The vertebrae to be instrumented is less than 12mm in height (based on the staple size)
4. One of the vertebrae to be instrumented in less than 20.5mm in width (base on smallest screw length)
5. One of the vertebrae to be instrumented is more than 44mm in width (base on longest screw length)
6. Non-idiopathic scoliosis
7. Non-ambulatory
8. Subject with clinical diagnosis of osteoporosis, osteopenia, osteomalacia, Paget's disease and metabolic bone disease
9. Prior thoracic surgery
10. Abnormal neurological status at baseline
11. Any condition or therapy that the investigator believes might pose a risk to the participant or make participation in the study not in the participant's best interest

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of device- &/or procedure-related SAEs | 12 months
  Rate of positively adjudicated device or procedure related serious adverse events including subsequent secondary surgical intervention and neurological events from baseline (preoperative) through 12 months
Change in Cobb angle measurement | 12 months
  The change in Cobb angle measurement from baseline (preoperative) to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Firoz Miyanji, Principal Investigator — BC Children's; Kevin Smit, Principal Investigator — CHEO
Locations (1):
- CHEO, Ottawa, Canada

IPD SHARING:
Plan to Share IPD: No